CLINICAL TRIAL: NCT07363720
Title: A Double-blind, Placebo-Controlled, Randomized Withdrawal Trial to Evaluate the Efficacy and Safety of TAK-861 for the Treatment of Narcolepsy With Cataplexy (Narcolepsy Type 1)
Brief Title: A Trial of TAK-861 for the Treatment of Narcolepsy With Cataplexy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-861-3003; 2024-519466-44-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Narcolepsy Type 1 (NT1); Narcolepsy With Cataplexy
Keywords: Drug Therapy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Double-blind RW Period: TAK-861 (Experimental): Participants on stable TAK 861 dose will receive the same dose of TAK-861 they were taking at the end of the OL treatment period, for up to 4 weeks in the double-blind RW period.
  Interventions: Drug: TAK-861
- Double-blind RW Period: Placebo (Placebo Comparator): Participants will receive TAK-861 matching-placebo, for up to 4 weeks in the double-blind RW period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-861 — TAK-861 tablets
  Arms: Double-blind RW Period: TAK-861
Drug: Placebo — TAK-861-matching placebo tablets
  Arms: Double-blind RW Period: Placebo

SUMMARY:
The main aim of this study is to assess how effective TAK-861 is for treating narcolepsy type 1 and if this effect is maintained over time. Participants will take TAK-861 for a few months and if they meet certain criteria, they will be randomly assigned (by chance, like flipping a coin) to continue taking TAK-861 or take placebo (fake medicine) for up to 4 weeks to see if their narcolepsy symptoms return.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-861. This study will look at how effective TAK-861 is for the treatment of narcolepsy type 1 and how well this effect is maintained over time. This study also evaluates how safe TAK-861 is and what adverse events may be associated with taking the drug and stopping the drug in participants with NT1.

The study will enroll approximately 88 participants. All participants will take TAK-861 during the open-label (OL) treatment period. Participants who meet certain criteria at the end of the OL Treatment Period will be randomized to one of two treatment groups for the up to 4-week double-blind randomized withdrawal (RW) Period. Participants will be randomized to one of the following treatment groups during the Double-blind RW Period:

1. TAK-861 (same dose participant was taking at the end of the OL Treatment Period)
2. Placebo

The randomized withdrawal period may last up to 4 weeks. Participants whose NT1 symptoms get worse during the RW period and whose Epworth Sleepiness Scale score rises above a certain score will stop the treatment and be invited to continue in a separate long term extension study. Participants who choose not to take part in the extension study will be followed-up for 4 weeks after their last dose of study drug. This multi-center trial will be conducted globally.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has a body mass index (BMI) within the range 18 to 40 kilograms per square meter (kg/m^2).
2. The participant has an International Classification of Sleep Disorders, Third Edition (ICSD-3) or International Classification of Sleep Disorders, Third Edition, Text Revision (ICSD-3-TR) diagnosis of NT1.
3. The participant is positive for the human leukocyte antigen (HLA) genotype Major Histocompatibility Complex, Class II, DQ Beta 1 (HLA-DQB1*06:02) or results from radioimmunoassay indicate the participant's CSF OX/hypocretin-1 concentration is ≤110 pg/mL (or less than one-third of the mean values obtained in normal participants within the same standardized assay).

Exclusion Criteria:

1. The participant has a current medical disorder, other than narcolepsy with cataplexy, associated with EDS.
2. The participant a) has a history of myocardial infarction, b) has a history of clinically significant hepatic disease, thyroid disease, coronary artery disease, cardiac rhythm abnormality or heart failure, or c) has any medical condition (such as unstable cardiovascular, pulmonary, renal or gastrointestinal disease.
3. The participant has current or recent (within 6 months) gastrointestinal disease that is expected to influence the absorption of drugs.
4. The participant has a history of cancer in the past 5 years.
5. The participant has a clinically significant history of head injury or head trauma.
6. The participant has a history of epilepsy, seizure, or convulsion (except for a single febrile seizure in childhood).
7. The participant has a history of cerebral ischemia, transient ischemic attack (less than 5 years from screening), intracranial aneurysm, or arteriovenous malformation.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Time to Loss of Response in the Epworth Sleepiness Scale (ESS) Score During the Up to 4-Week RW Period | Up to 4-week RW period
  The ESS provides individuals with 8 different situations of daily life and asks them how likely they are to fall asleep in those situations (scored 0 to 3) and to try to imagine their likelihood of dozing even if they have not actually been in the identical situation; the scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within normal range.

SECONDARY OUTCOMES:
Change From the End of the OL Treatment Period to Week 2 of the RW Period on the Maintenance of Wakefulness Test (MWT) | From the end of the OL treatment period (Week 16) to Week 2 of the RW period (Week 18)
  The MWT evaluates a person's ability to remain awake under soporific conditions for a defined period of time. Because there is no biological measure of wakefulness, wakefulness is measured indirectly by the inability or delayed tendency to fall asleep. This tendency to fall asleep is measured via electroencephalography (EEG)-derived sleep latency in the MWT. The MWT consists of four 40-minute sessions. Sleep latency in each wake trial will be recorded. Participants will be required to stay awake in between the 4 sessions.
Weekly Cataplexy Rate (WCR) at Week 2 of the RW Period | Week 2 of the RW period
Change from the End of the OL Treatment Period to Week 2 of the RW Period in Mean Number of Lapses on the Psychomotor Vigilance Test (PVT) | From the end of the OL treatment period (Week 16) to Week 2 of the RW period (Week 18)
  The PVT is a simple reaction performance task with a duration of 10 minutes that aims to measure sustained attention.
Number of Participants Reporting Much or Very Much Worse in Patient Global Impression of Change (PGI-C) Score at Week 2 of the RW Period | Week 2 of the RW period
  The PGI-C is a participant self-rated scale to assess improvement in daytime sleepiness and overall narcolepsy symptoms. It measures change due to treatment relative to baseline on a 7-point scale ranging from a score of 1 ("very much improved") to score of 7 ("very much worse").
Change from the End of the OL Treatment Period to Week 2 of the RW Period in Narcolepsy Severity Scale for Clinical Trials (NSS-CT) Total Score | From the end of the OL treatment period (Week 16) to Week 2 of the RW period (Week 18)
  The NSS-CT is a 15-item self-administered questionnaire assesses the severity and consequences of the 5 major narcolepsy symptoms such as daytime sleepiness, cataplexy, hallucinations, sleep paralysis, and disturbed night-time sleep (DNS) with a total score range of 0 to 57 (sum of 6 items that assess symptoms severity are rated using a six-point Likert scale [0-5] and 9 items that describe the symptom effect on daily life are rated using a four-point Likert scale [0-3]. Higher total scores mean a worse outcome.
Change from the End of the OL Treatment Period to Week 2 of the RW Period in Functional Impacts of Narcolepsy Instrument (FINI) Domain Scores | From the end of the OL treatment period (Week 16) to Week 2 of the RW period (Week 18)
  The FINI measures the functional impacts of narcolepsy across 6 domains. Each domain is scored from 0 to 4, where 0 indicates the best health and 4 the worst.
Change from the End of the OL Treatment Period to Week 2 of the RW Period in Number of Correct Responses on the International Digit Symbol Substitution Test-symbols (iDSST-s) | From the end of the OL treatment period (Week 16) to Week 2 of the RW period (Week 18)
  The iDSST-s is a processing speed test that is based on the pre-existing pencil and paper version of the Digit Symbol Substitution Test. The participants are presented with a legend that defines 9 symbols, with each symbol corresponding to a digit from 1 to 9. The participant is then presented with a conveyer belt in the middle of the screen that displays a series of empty boxes labelled with a number. The participant must select the symbol that corresponds to the number of a given highlighted box from symbol options presented at the bottom of the screen. The participant must try to place as many correct symbols in the boxes as possible over the duration of the test.
Number of Participants With At Least One Treatment-Emergent Adverse Event (TEAE) | From Screening to End of study (approximately 31 weeks)
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/